CLINICAL TRIAL: NCT01738802
Title: The Effects of Micronutrients in Combination With Usual Care in Type 2 Diabetes
Acronym: PMC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Alicia L. Warnock, Director, Diabetes Institute, Walter Reed National Military Medical Center
Allocation: Randomized | Model: Single Group | Masking: Triple
Other Study IDs: 361813
Record Dates: First submitted 2012-07-19; First posted 2012-11-30 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes; carotid intima medial thickness; micronutrient; anti-oxidant
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Antioxidants; Micronutrients

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Anti-oxidant and micronutrient (Experimental): This group will take the anti-oxidant and micronutrient supplement.
  Interventions: Dietary Supplement: Anti-oxidant and micronutrient
- Placebo (Placebo Comparator): This group will take the placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: Anti-oxidant and micronutrient — This group will be randomized to take the anti-oxidant and micronutrient supplement.
  Arms: Anti-oxidant and micronutrient
Drug: Placebo — This group will take a placebo.
  Arms: Placebo

SUMMARY:
This study is evaluating the impact of antioxidant supplements on blood sugar control and cardiovascular risk factors in adults over the age of 50 with at 3 months of Type 2 diabetes. The investigators hypothesize that daily supplementation with a multiple micronutrient formulation containing dietary and endogenous antioxidants in combination with usual care will reduce markers of oxidative stress and inflammation in Type 2 diabetes.

DETAILED DESCRIPTION:
This study is evaluating the impact of an antioxidant and micronutrient supplement on markers of oxidative stress and inflammation as well as on blood sugar control in adults over the age of 50 who have had Type 2 diabetes for at least 3 months. The purpose of this study is to see if these antioxidants reduce the oxidative and inflammatory state seen in patients with Type 2 diabetes as well as whether or not they make it easier to control blood sugar, affect the number and dosage of diabetic medications, and/or reduce the risk factors involved in long-term diabetes related complications such as in lipid profile and carotid intima-media thickness (CIMT).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a diagnosis of Type 2 diabetes of at least three months duration
2. 50 years of age or older
3. Stable medical status (e.g., no myocardial infarction, stroke, major surgery, or major mental illness during the previous six months)
4. Not taking or not expected to be taking any oral glucocorticoids (except for replacement therapy for those with adrenal insufficiency), amphetamines, anabolic, or weight-reducing agents during the course of the study
5. Not receiving chemotherapy or immunosuppressive therapy
6. Military healthcare beneficiary

Exclusion Criteria:

1. Patients with Type 1 diabetes or those with Type 2 diabetes of less than 3 months duration.
2. Inability to communicate in written and spoken English
3. Organ (kidney, pancreas, liver) transplant recipients
4. Individuals who are not likely to return for the follow-up because they or their sponsors are likely to have a permanent change of station or termination of service before completion of the protocol
5. Pregnancy (Women who are pre-menopausal will be informed that pregnancy must be ruled out by a serum HCG test if they would like to be considered for participation in the study. Women who have had a hysterectomy or have not had a menstrual period for at least one year prior to consent will be considered post-menopausal and will not require a serum pregnancy test).
6. Patients who are routinely taking more than 81 mg aspirin (ASA)/day or who are using ASA or ASA-containing products to manage a chronic condition.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2012-01; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Change in the markers of oxidative stress and inflammation | baseline, 6, and 12 months
  Determining a difference between the control and experimental groups in the following markers of 1) oxidative stress: 9-Malondialdehyde (MDA) in plasma, 3-Nitrotyrosine in plasma, and Urinary levels of F2-isoprostane and 8 hydroxy,deoxyguanosine; and 2) inflammation: GM-CSF, IFN-γ, IL-1β, IL-2, L-4, IL-5, IL-6, IL-10, IL-12 (p40/p70), TNF-α.

SECONDARY OUTCOMES:
Change in CIMT | Baseline, 6 and 12 months
  Determine if a difference exists in CIMT measurements between the control and experimental groups.
Change in medications | Baseline, 3, 6, 9, and 12 months
  Compare the experimental and control groups to determine if medication use has changed over the course of the study.
Change in lipid profile | baseline, 3, 6, 9, and 12 months
  Compare the control and experimental groups to determine differences in lipid profile over time.
Hemoglobin A1c | baseline, 3, 6, 9, and 12 months
  Determine the difference in quarterly A1c measurements between the experimental and control groups over the course of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Vigersky, MD, Principal Investigator — WRNMMC
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States